## STATISTICAL PLAN

| Time-based R | Register and | Analysis o | of COPD En | dpoints | (TRACE). |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

NCT number: NCT03485690

Date: February 2<sup>nd</sup>, 2018

## Scientific committee:

Jose Luis Lopez-Campos Bodineau

Laura Carrasco Hernández

María Abad Arranz

Eduardo Márquez Martín

Carmen Calero Acuña

Francisco Ortega Ruiz

## Institutions:

- Centro de investigación biomédica en red de enfermedades respiratorias (CIBERES).
   Instituto de Salud Carlos III, Madrid Spain
- (2) Unidad Médico-Quirúrgica de Enfermedades Respiratorias, Instituto de Biomedicina de Sevilla (IBiS), Hospital Universitario Virgen del Rocío/Universidad de Sevilla, Seville,

  Spain

## Statistical plan

The data will be analyzed using the software IBM SPSS Statistics (IBM corporation, Armonk, New York). For the description of the variables, centralization and dispersion estimators appropriate to the nature of each variable and its distribution will be used. The differences between baseline patient types will be analyzed using the Student's t test for independent data (after checking the equality of the variances with the Levene test) or using the Chi-square test (with Fisher's correction if applicable) for qualitative variables. Follow-up studies will be done using the Student's t test for paired data or with the McNemar test for categorical variables. Potential associations found in this bivariate analysis will be further evaluated via a multivariate study depending on the nature of the analysis. Accordingly, the calculation of the relative risk of future events will be adjusted from multiple regression models. Survival analysis will be carried out by Kaplan-Meier curves with log-rank test to assess differences between potential patient groups. Potential associations will be further explored by Cox proportional hazards regression analysis. The level of statistical significance is set at 0.05.